CLINICAL TRIAL: NCT01817036
Title: Knowledge Innovation Project of CAS - Genetic and Nutritional Association Studies on Metabolism-related Diseases in Chinese Population -- Vitamin D Intervention Study：A Pilot Study
Brief Title: Vitamin D Intervention Trial in Healthy Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSCX2-EW-R-10-VD
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; deficiency; dose response
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Placebo (Placebo Comparator): 5 placebo pills per day, 16 weeks
  Interventions: Dietary Supplement: Placebo
- 400 IU (Experimental): (4 placebo pills + 1 vitamin D pill) per day, 16 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D
- 800 IU (Experimental): (3 placebo pills + 2 vitamin D pills) per day, 16 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D
- 1200 IU (Experimental): (2 placebo pills + 3 vitamin D pills) per day, 16 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D
- 2000 IU (Experimental): 5 vitamin D pills per day, 16 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Placebo — placebo
  Arms: 1200 IU; 400 IU; 800 IU; Placebo
Dietary Supplement: Vitamin D — 400 IU vitamin D per pill
  Arms: 1200 IU; 2000 IU; 400 IU; 800 IU

SUMMARY:
To determine the dose-response between the doses of vitamin D3 supplements and raised serum levels of 25(OH)D and also the dose of vitamin D3 required to achieve circulating 25(OH)D ≥ 75 nmol/L;

DETAILED DESCRIPTION:
Recent epidemiological studies suggested that serum 25-hydroxyvitamin D [25(OH)D] concentration ≥75 nmol/L appeared to be optimal for preventing cardiometabolic diseases and improving bone health. To achieve this goal, a daily intake of 1000 IU or equivalent amount from other sources, is needed, which is twice as much as the RDA recommended by Chinese Nutrition Society. Meanwhile,epidemiological evidences show that large proportions of Chinese may suffer vitamin D insufficiency or deficiency whereas the current RDA in China might be too low to provide adequate vitamin D for people's health.

In order to fill up this gap, therefore, it is essential to determine the dose-response between the doses of vitamin D3 supplements and raised serum levels of 25(OH)D and also the dose of vitamin D3 required to achieve circulating 25(OH)D ≥ 75 nmol/L.Ultimately, the current study will provide important evidence for establishing optimal vitamin D requirement for Chinese people

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-45 years. with vitamin D deficiency (25(OH)D < 50 nmol/l)

Exclusion Criteria:

* BMI < 18.5 kg/m2, or BMI ≥ 25 kg/m2
* Total intake of calcium from diet or supplements >1200mg/d, or fasting serum calcium level ≥2.75 mmol/l
* Participating in other clinical studies within previous 3 months
* Taking vitamin D supplements within previous 3 months
* Using medications that may affect vitamin D metabolism in previous 3 months;
* Concomitant with clinical conditions, like liver dysfunction (serum alanine transaminase (ALT) ≥40 U/L; and/or aspartate transaminase (AST) ≥40 U/L; Glutamyl transpeptidase （GGT）≥50 U/L; serum creatinine < 50 or > 120 µmol/L; urea nitrogen (UN) < 7 or > 18 mg/dl, and/or urine acid <90 or >420 µmol/L; which may affect vitamin D metabolism;
* History of drug or alcohol abuse (>40 g/d)
* Women during pregnancy or lactation
* Individuals with mental disorders or current use of antidepressants, the conditions which may affect him or her understanding and unwillingness to the intervention;
* Having clinically diagnosed AIDS, hepatitis A, hepatitis B, tuberculosis and other infectious diseases.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D | 16 weeks
  Serum 25(OH)D concentration will be assayed by utilizing a liquid chromatography-mass spectrometry (LC-MS) method

SECONDARY OUTCOMES:
alanine aminotransferase（ALT) | 16 weeks
  Serum ALT will be measured by an Automatic biochemical analyzer
aspartate aminotransferase(AST) | 16 weeks
  Serum AST will be measured by an Automatic biochemical analyzer;
glutamyl transpeptidase（GGT） | 16 weeks
  Serum GGT will be measured by an Automatic biochemical analyzer
creatinine | 16 weeks
  creatinine will be measured by an Automatic biochemical analyzer
uric acid | 16 weeks
  Serum uric acid will be measured by an Automatic biochemical analyzer
urea nitrogen | 16 weeks
  Serum urea nitrogen will be measured by an Automatic biochemical analyzer
calcium | 16 weeks
  Serum calcium will be measured by an Automatic biochemical analyzer.
phosphate | 16 weeks
  Serum phosphate will be measured by an Automatic biochemical analyzer.
parathyroid hormone（PTH） | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences, Shanghai, Shanghai Municipality, China